CLINICAL TRIAL: NCT06064578
Title: The Ukrainian Student Problem Solving Project: A Randomized Effectiveness Trial of a Brief, Digital Problem Solving Intervention for Youth
Brief Title: The Ukrainian Student Problem Solving Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard University (Other)
Collaborators: King's College London (Other)
Responsible Party: Principal Investigator, John Weisz, Professor, Harvard University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB23-0975
Record Dates: First submitted 2023-09-26; First posted 2023-10-03 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Trauma; Anxiety; Depression; Child Behavior
MeSH Terms: conditions — Wounds and Injuries; Anxiety Disorders; Depression; Child Behavior

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive the intervention condition (Project SOLVE) immediately or after three months. Participants in the delayed SOLVE condition will complete a typical school activity instead (i.e., treatment as usual). All participants will complete follow-up measures online at baseline, immediately after receiving the intervention, and 1-, 3, 4-, and 6-months after baseline.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Assessments will be completed independently by participants online. Investigators will be blinded to condition throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Project SOLVE (Experimental): Project SOLVE is a ~30-minute self-guided digital intervention designed to teach children and adolescents how to set goals and solve problems systematically. Specifically, Project SOLVE is based on problem solving, a core component of cognitive behavioral therapy, a gold standard treatment for internalizing disorders. Project SOLVE uses vignettes, interactive activities, and engaging graphics to teach youth a systematic strategy for solving problems. Project SOLVE was previously found to be effective in reducing mental health symptoms among American children (https://link.springer.com/article/10.1007/s12310-023-09598-7).
  Interventions: Behavioral: Project SOLVE
- Delayed Receipt of Project SOLVE Control Condition (Other): No intervention for first three months; will receive SOLVE after 3-months and become a second-wave intervention condition.
  Interventions: Behavioral: Project SOLVE

INTERVENTIONS:
Behavioral: Project SOLVE — Project SOLVE is a ~30-minute self-guided digital intervention designed to teach children and adolescents how to set goals and solve problems systematically. Specifically, Project SOLVE is based on problem solving, a core component of cognitive behavioral therapy, a gold standard treatment for internalizing disorders. Project SOLVE uses vignettes, interactive activities, and engaging graphics to teach youth a systematic strategy for solving problems. Project SOLVE was previously found to be effective in reducing mental health symptoms among American children (https://link.springer.com/article/10.1007/s12310-023-09598-7).

SUMMARY:
The purpose of this study is to test the effectiveness of a universal, digital, single-session intervention for youth mental health, functioning, and well-being. The investigators will be providing access to a brief online program (Project SOLVE) for students as part of the school curriculum. Ukrainian students living in Poland will be randomly assigned to receive Project SOLVE either immediately or after 3 months. The program is designed to help students manage stress and reach their academic and personal goals by teaching them how to solve problems systematically. The investigators would like to evaluate the effectiveness of this intervention in improving students' mental health and well-being.

DETAILED DESCRIPTION:
Half of all Ukraine war refugees are children; more than one million are in Poland, coping with multiple traumas (e.g., war, evacuation, family separation) that threaten their mental health (MH). Since meetings in Warsaw in summer 2022, PI Weisz has worked with child mental health researchers and clinicians from Ukraine and 5 other countries (the GROW consortium) and with staff of Ukrainian-language schools for displaced children to plan psychological support for the children. It is clear that Ukrainian-language digital MH interventions teaching empirically supported skills are the optimum scalable form of early psychological support, given the massive number of Ukrainian children, their dispersion to diverse countries, the dearth of professional clinicians, and the ready accessibility of digital devices. They require no professional training or funding, and are easily implemented via digital devices used in virtually all schools.

Primary child MH problems identified by research reviews and the school staff include anxiety, difficulty calming and regulating negative emotions, and diverse interpersonal and adaptation problems. The BDI, Project SOLVE helps children identify problems they can solve, and use 5 simple steps to solve them. This 30-40-minute BDI, refined via student and school staff feedback, highly rated by children, has each been accessed >750 times in the U.S. and Canada; SOLVE was found effective in a recent RCT.

Using a randomized controlled design, the investigators will test Project SOLVE with students in partner schools. Students will be randomized to receive SOLVE immediately or three months later, with students assigned to the delayed condition participating in a typical school activity instead. Using this design, the investigators can test the intervention and ensure that no student is denied access. Students will complete MH, wellbeing, and BDI-skills (i.e., mechanism of change) measures at baseline, 1-, 3-, 4-, and 6-months after baseline. Students will be randomized 50/50 to receive Project SOLVE immediately or in three months. Parents will complete parent forms of all the measures at the same time points.

ELIGIBILITY:
Inclusion Criteria:

* Youth in grades 5+ at partnering schools for Ukrainian children
* Youth and at least one guardian consent to adolescent participation in study
* Youth reads Ukrainian well enough to effectively complete the digital programs
* Youth has access to a digital device

Exclusion Criteria:

* Youth does not have access to a digital device
* Youth has an intellectual disability that precludes comprehension of the program content

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 778 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Behavior and Feelings Survey (Internalizing Subscale; Students and Caregivers) | Assessed at baseline, 1-month, 3-month, 4-month, and 6-month follow-ups
  Trajectories of self-reported symptoms of anxiety and depression from the 6-item (each item rated on a 0-4 scale, with higher ratings indicating more symptoms) Internalizing subscale of the Behavior and Feelings Survey. Total scores range from 0 to 24, with higher scores indicating more symptoms.
Perceived Program Acceptability and Helpfulness (Students Only) | Assessed immediately post-intervention
  Post-intervention feedback on the program's perceived acceptability and helpfulness as measured via a 7-item scale, with each item rated on a 1-5 scale, with higher scores indicating greater acceptability and helpfulness.

SECONDARY OUTCOMES:
Change in Behavior and Feelings Survey (Externalizing Subscale; Students and Caregivers) | Assessed at baseline, 1-month, 3-month, 4-month, and 6-month follow-ups
  Trajectories of self-reported misbehavior from the 6-item (each item rated on a 0-4 scale, with higher ratings indicating more symptoms) Externalizing subscale of the Behavior and Feelings Survey. Total scores range from 0 to 24, with higher scores indicating more symptoms.
Student Problem-Solving Mechanisms of Change Questions (Students and Caregivers) | Assessed at baseline, 1-month, 3-month, 4-month, and 6-month follow-ups
  Assessed via a novel 3-item measure (0-10 scale) evaluating participants' problem-solving skills. Specific items include:
  * When I have a problem with another kid, I can solve it.
  * When I have a problem at home, I can solve it.
  * When I have a problem at school, I can solve it
Treatment Expectancy Questions (Students Only) | Assessed immediately pre-intervention
  Treatment expectations will be assessed at pre-intervention via a novel 4-item measure (0-10 scale) evaluating participants' expectations of intervention effects.
Peabody Treatment Progress Battery's Life Satisfaction Scale (Students and Caregivers) | Assessed at baseline, 1-month, 3-month, 4-month, and 6-month follow-ups
  Assessed via the Peabody Treatment Progress Battery's Life Satisfaction Scale. Items are rated on a scale from 1 (very dissatisfied) to 5 (very satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Harvard University, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Analytic code will be made available upon publication of trial results. Study protocol and statistical plan are available on Open Science Framework.
Supporting Information: Analytic Code
Time Frame: To be shared on OSF once data collection and analyses are complete.
URL: https://osf.io/u495j